CLINICAL TRIAL: NCT06988553
Title: A Phase Ib, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AZD5004 in Chinese Participants With Overweight/Obesity With or Without Type 2 Diabetes Mellitus
Brief Title: A Phase Ib Study of AZD5004 in Chinese Participants With Overweight/Obesity With or Without Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eccogene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D7260C00005
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-08

CONDITIONS: Obesity or Overweight; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AZD5004 (Experimental): Participants will receive AZD5004 orally.
  Interventions: Drug: AZD5004
- Placebo (Placebo Comparator): Participants will receive Placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5004 — AZD5004 will be administered as an oral tablet once daily.
  Arms: AZD5004
Drug: Placebo — Placebo will be administered as an oral tablet once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and PK of AZD5004 compared with placebo in Chinese participants with overweight/obesity with or without T2DM.

DETAILED DESCRIPTION:
This is a Phase Ib, randomized, parallel-group, double-blind, placebo-controlled, multicentre, 2-arm treatment study to investigate the safety, tolerability, and PK of AZD5004 compared with placebo in Chinese male and female participants aged 18 to 74 years, who are overweight/obese with or without T2DM. The primary endpoints are incidence of AEs, SAEs, DAEs, death, AESIs, laboratory parameters, 12-lead ECG, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 74 years inclusive at the time of signing the informed consent.
* Stable self-reported body weight for 3 months prior to Screening.

Inclusion Criteria for Cohort A:

- 27 kg/m2 ≤ BMI ≤ 35 kg/m2 and weigh at least 60 kg at Screening.

Inclusion Criteria for Cohort B:

* Diagnosed with T2DM for at least 6 months prior to signing the informed consent.
* HbA1c value at Screening of ≥ 7.0% and ≤ 10.5%
* BMI of ≥ 24 kg/m2 at the Screening Visit.

Exclusion Criteria:

* History of, or any existing condition that influence the participant's ability to participate or affect the interpretation of the results of the study.
* Known clinically significant gastric emptying abnormality.
* Significant hepatic disease.
* Abnormal renal function.
* History of acute pancreatitis and chronic pancreatitis, gallstones.
* Uncontrolled thyroid disease.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), serious adverse events (SAEs), adverse event leading to the discontinuation of study intervention (DAEs), death, and Adverse events of special interest (AESIs) | From baseline to week 16.
  To evaluate the safety and tolerability of AZD5004 compared with placebo.

SECONDARY OUTCOMES:
AZD5004 concentrations in plasma | Week 16.
  To characterize the PK profile of AZD5004 following repeated administration.
Area under the concentration-time curve over a dosing interval (AUCtau) | Week 16.
  To characterize the PK profile of AZD5004 following repeated administration.
Maximum Observed Plasma Concentration (Cmax) | Week 16.
  To characterize the PK profile of AZD5004 following repeated administration.
Half-Life (t1/2) | Week 16.
  To characterize the PK profile of AZD5004 following repeated administration.
Time of Occurrence of Maximum Plasma Concentration (tmax) | Week 16.
  To characterize the PK profile of AZD5004 following repeated administration.
Trough concentration (Ctrough) | Week 16.
  To characterize the PK profile of AZD5004 following repeated administration.

CONTACTS AND LOCATIONS:
Overall Officials: Eccogene, Study Director — Eccogene Clinical Trials
Locations (6):
- China (6):
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Fourth Affiliated Hospital of Harbin Medical University, Ha’erbin
  - The Second People's Hospital of Hefei, Hefei
  - Jinan Central Hospital, Jinan
  - Shanghai Pudong New District People's Hospital, Shanghai
  - General Hospital of Tianjin Medical University, Tianjin

IPD SHARING:
Plan to Share IPD: No